CLINICAL TRIAL: NCT02767492
Title: A Double-blind, Randomized Study Comparing Steroid Injection and BioDRestore for Patients With Knee Osteoarthritis
Brief Title: Steroid Injection vs. BioDRestore for Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hawkins Foundation (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00048698
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioDRestore™ (Experimental): BioDRestore™ Elemental Tissue Matrix is a morselized, flowable tissue allograft derived from amniotic tissues. 2cc will be injected in the knee joint.
  Interventions: Device: BioD Restore
- Corticosteroid (Active Comparator): Kenalog (40 mg of 40 mg/ml) will be the steroid utilized as the active comparator to be injected in the knee joint.
  Interventions: Drug: Kenalog

INTERVENTIONS:
Device: BioD Restore — Investigational product, BioD Restore, will be injected into the articular space of the knee.
  Arms: BioDRestore™
Drug: Kenalog — Active comparator, Kenalog steroid, will be injected into the articular space of the knee.
  Arms: Corticosteroid

SUMMARY:
This study will include patients who are diagnosed with knee OA and are recommended for a knee injection. Study subjects will be randomized to receive either the standard of care knee injection (steroid) or amniotic tissue injection (BioDRestore). Study subjects will be asked for permission for a baseline knee aspiration prior to the knee injection. At 6 months post-injection, knee aspirations will be taken and sent for analysis. Study subjects will be followed for 1 year post-injection to include range of motion measurements and patient-reported pain/functional outcome measurements. X-rays will also be taken at the 1-year post-injection appointment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 80 years.
* Willing and able to give voluntary informed consent to participate in this investigation.
* Patient presents with knee osteoarthritis and Kellgren Lawrence grade 2-4 (OA diagnosed and confirmed by treating physician using standing x-ray).
* Candidate for intra-articular knee injection.
* BMI < 40

Exclusion Criteria:

* Patients who have received intra-articular injection(s) in the last 3 months.
* Patients who have undergone arthroscopic surgery on the study knee in the past year.
* Patients who have undergone arthroplasty on the study knee.
* Ligament instability
* Diabetes (Type 1 or II)
* Inflammatory arthropathies.
* Fibromyalgia or chronic fatigue syndrome.
* Female patient who is pregnant or nursing.
* Chronic use of narcotics.
* Any other reason (in the judgment of the investigator).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Siffri, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Health System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pill SG, Ahearn B, Tokish JM, Cook C, Siffri PJ, Mercuri JJ, Burnikel B, Cassas KJ, Wyland DJ, Sawvell E, Wright N, Hutchinson J, Bynarowicz T, Adams KJ, Kissenberth MJ. Amniotic Tissue Injections Are an Effective Alternative to Corticosteroid Injections for Pain Relief and Function in Patients With Severe Knee Osteoarthritis: A Double-Blind, Randomized, Prospective Study. J Am Acad Orthop Surg Glob Res Rev. 2025 Jan 9;9(1):e23.00276. doi: 10.5435/JAAOSGlobal-D-23-00276. eCollection 2025 Jan 1. PMID 39813395

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BioDRestore™ | Corticosteroid
Started | 45 | 45
Completed | 35 | 35
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BioDRestore™ | Corticosteroid | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.86 (8.98) | 64.03 (8.92) | 62.92 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 17 | 20 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 44 | 44 | 88
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 43 | 42 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Score
Description: Patient reported level of pain on a scale of 0-10, with 10 being extreme pain and 0 being no pain.
Time Frame: Surgery through 12 months post-op/
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioDRestore™ | Corticosteroid
Number analyzed (Participants) | 35 | 35
score on a scale | 2.49 (2.41) | 3.25 (2.82)

2. Primary Outcome: Veterans Rand 12 Item Health Survey
Description: Patient reported quality of life. Score contains a physical component and mental component score. Both scales are continuous and values range from 0 to 70, with higher scoring indicating higher physical and mental component scores
Time Frame: Sugery to 12 months post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioDRestore™ | Corticosteroid
Number analyzed (Participants) | 35 | 35
score on a scale | 56.95 (9.84) | 58.01 (7.49)

3. Primary Outcome: Lysholm Knee Score
Description: Patient reported knee function scores on a scale of 0-100, with 100 being a excellent outcome indicating no symptoms.
Time Frame: Surgery to 12 months post-op.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioDRestore™ | Corticosteroid
Number analyzed (Participants) | 35 | 35
score on a scale | 75.26 (17.75) | 61.00 (22.00)

4. Primary Outcome: Single Alpha Numeric Evaluation (SANE)
Description: Percentage of normal for affected knee between 0 to 100, with 100 being a perfectly "normal" knee and 0 being a completely "abnormal" knee.
Time Frame: Surgery to 12 months post-op.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioDRestore™ | Corticosteroid
Number analyzed (Participants) | 35 | 35
score on a scale | 66.14 (23.27) | 60.49 (25.37)

5. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: Knee outcome measure assessed via Knee Injury and Osteoarthritis Outcome Score (KOOS) on a scale of 0 to 100. The higher score of 100 indicates a fully functional knee without knee pain or problems.
Time Frame: Surgery to 12 months post op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BioDRestore™ | Corticosteroid
Number analyzed (Participants) | 35 | 35
score on a scale | 64.10 (21.23) | 55.67 (22.23)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | BioDRestore™ | Corticosteroid
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT02767492/Prot_SAP_000.pdf